CLINICAL TRIAL: NCT00041743
Title: Treatment of Binge Eating Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: Crow (completed)
Record Dates: First submitted 2002-07-16; First posted 2002-07-17 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder

INTERVENTIONS:
Behavioral: Group Cognitive Behavioral Therapy

SUMMARY:
This is a study examining the use of different degrees of therapist involvement in the treatment of Binge Eating Disorder. The study will examine both which approaches work best for decreasing symptoms and which are most cost-effective.

ELIGIBILITY:
* Binge Eating Disorder
* Age 18-65, Male or Female
* Not Currently receiving psychotherapy
* Not currently in Formal weight loss treatment
* No current unstable medical problems
* No history of Bipolar illness or Schizophrenia
* Overweight or Obese (body mass index 25-45)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-07; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott J Crow, MD, Principal Investigator — Universtiy of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Pacanowski CR, Mason TB, Crosby RD, Mitchell JE, Crow SJ, Wonderlich SA, Peterson CB. Weight Change over the Course of Binge Eating Disorder Treatment: Relationship to Binge Episodes and Psychological Factors. Obesity (Silver Spring). 2018 May;26(5):838-844. doi: 10.1002/oby.22149. Epub 2018 Mar 13. PMID 29533531
- [Derived] Pisetsky EM, Durkin NE, Crosby RD, Berg KC, Mitchell JE, Crow SJ, Wonderlich SA, Peterson CB. Examination of early group dynamics and treatment outcome in a randomized controlled trial of group cognitive behavior therapy for binge eating disorder. Behav Res Ther. 2015 Oct;73:74-8. doi: 10.1016/j.brat.2015.07.013. Epub 2015 Jul 31. PMID 26264648
- [Derived] Peterson CB, Mitchell JE, Crow SJ, Crosby RD, Wonderlich SA. The efficacy of self-help group treatment and therapist-led group treatment for binge eating disorder. Am J Psychiatry. 2009 Dec;166(12):1347-54. doi: 10.1176/appi.ajp.2009.09030345. Epub 2009 Nov 2. PMID 19884223